CLINICAL TRIAL: NCT04047810
Title: A Pilot Study to Evaluate the Safety and Feasibility of Mesenchymal Stem Cells in the Treatment of Subjects With Advance Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Mesenchymal Stem Cells in the Treatment of Subjects With Advance Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jorge M Mallea, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-007748
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects with Advanced Chronic Obstructive Pulmonary Disease (Experimental): Subjects diagnosed with severe or very severe COPD will be infused intravenously with Mesenchymal Stem Cells (MSC)
  Interventions: Biological: Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Mesenchymal Stem Cells — 0.5- 2 million cells/kg, intravenously once

SUMMARY:
Researchers are trying to understand the effects of mesenchymal stem cells therapy in subjects with advance chronic obstructive pulmonary disease

ELIGIBILITY:
Inclusion Criteria

* Age range: at least 18 years of age
* Gender: Male or female
* Target disease or condition: Subjects with advance COPD
* Subject must have a post-bronchodilator FEV1/FVC ratio of less than 0.7
* Subject must have a post-bronchodilator FEV1percent predicted value between 20% and 49%.
* Subject must have a total lung capacity (TLC) percent predicted of 80% or more
* Subject must be an ex-smoker, with a cigarette smoking history of ≥ 10 pack-years.
* Subject must have abstained from nicotine products for at least six months prior to enrollment in the study.
* Subjects must score at least 2 in the modified Medical Research Council (mMRC)
* Subjects must have had an exacerbation of COPD within the last 12 months prior to enrollment in the study. An acute exacerbation of COPD is defined as a respiratory event requiring the use of antibiotics or systemic steroids or both.
* Informed consent form (ICF): Each patient will be required to sign an IRB approved ICF. Only subjects who have signed the ICF will be enrolled into the study. The ICF will include elements required by Mayo IRB and FDA in US 21CFR50.
* Subject must have a calculated creatinine clearance of greater than 30 ml/min.
* Subject must be available for all specified assessments at the study site through the completion of the study.
* Subject must provide written ICF and authorization for use of and disclosure of PHI.
* Subjects must have oxyhemoglobin saturation on room air at rest equal or greater than 88%.

Exclusion Criteria

* Patients with clinically significant illness with manifestations of significant organ dysfunction which in the judgment of the PI or co-investigator would render the study subject unlikely to tolerate the MSC infusion or complete the study
* Subject has been diagnosed with a pulmonary disease other than COPD (e.g. asthma, pulmonary fibrosis, sarcoidosis, pulmonary hypertension, bronchiolitis, interstitial lung disease)
* Subject has been diagnosed with α1-Antitrypsin deficiency
* Subject has a body mass index greater than 35 or less than 16
* Subject has or has had an active infection requiring systemic antibiotics within 12 weeks on enrollment in the study
* Subject has had exacerbation of COPD requiring hospitalization within 12 weeks of enrollment in the study.
* Subject has initiated pulmonary rehabilitation within 12 weeks of enrollment in the study
* Subject uses or used prednisone (or equivalent dose of another corticosteroid) within 12 weeks of enrollment in the study
* Subject has evidence or history of malignancy
* Subject has evidence or history of autoimmune disorders independent of COPD
* Subject is pregnant or breast-feeding
* Subject has a history of HIV, Hepatitis B and/or Hepatitis C
* Subject has evidence of liver dysfunction manifested as alkaline phosphatase greater than 345 u/L, total bilirubin greater than 1.65 mg/dL, ALT greater than 275 units/L and/or AST great than 240 units/L.
* Subject has evidence of significant cardiac dysfunction, e.g. acute myocardial infarction within 3 months of screening, patients with the diagnosis of unstable angina. Patients with the diagnosis of "Cor pulmonale", uncontrolled tachyarrhythmia or bradyarrhythmia, atrial fibrillation or atrial flutter, history of insertion of pacemaker or implantable cardioverter-defibrillator, patient with clinical diagnose of heart failure with preserved or reduced ejection fraction and patients with a history of congenital heart disease.
* Subjects with pulmonary lobectomy or lung volume reduction surgery or lung transplantation.
* Subjects with clinically significant bronchiectasis.
* Subject received an experimental therapy (drug or biologic) for any indication within 12 months of the study enrollment
* Subject is unable to complete all the testing required for the study
* Subjects who are on immunosuppressive medications.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Adverse Events | One hour post completion of infusion
  Number of subjects to tolerate IV infusion of Mesenchymal Stem Cells (MSC) without acute clinical or physiological deterioration

CONTACTS AND LOCATIONS:
Overall Officials: Jorge M Mallea, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials